CLINICAL TRIAL: NCT03685292
Title: "Fraud Case Study" - The Tone At The Top and What Constitutes Criminal Behavior.
Brief Title: Behavioral Studies and Practices
Acronym: BSPJ
Status: Completed | Type: Observational
Sponsor: Brian Bolden (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Brian Bolden, Student, Foundation of iAesthetics and Neurobiology
Organization: Foundation of iAesthetics and Neurobiology (Other)
Other Study IDs: Behavioral Studies Journal; 0037 (Registry Identifier: Southern University and A&M Colleges)
Record Dates: First submitted 2018-07-19; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-07

CONDITIONS: Behavioral
MeSH Terms: conditions — Behavior | interventions — Behavior Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Group A: Subject(s): A Subgroup
  Interventions: Behavioral: Behavioral Advisory System; Drug: Behavioral Treatment; Device: Behavioral Division
- Group B: Subject(s): B Subgroup
  Interventions: Behavioral: Behavioral Advisory System; Drug: Behavioral Treatment; Device: Behavioral Division
- Group C: Subject(s): C Sub Group
  Interventions: Behavioral: Behavioral Advisory System; Drug: Behavioral Treatment; Device: Behavioral Division

INTERVENTIONS:
Behavioral: Behavioral Advisory System — Support and training to help increase throughput while promoting upstanding stature and reproducibility in behavioral testing using cutting edge methodologies.
  Other Names: Triple Helix Methodology System
Drug: Behavioral Treatment — This study addressed the efficacy of cognitive-behavioral therapy (CBT) treatment.
Device: Behavioral Division — This study is relative to minimal contact control (MCC).

SUMMARY:
The focus of this study is to evaluate whether a new fraud material will be suitable for a technological device and or software. ***For consultation purposes only.***

ELIGIBILITY:
Inclusion Criteria:

* College Student

Exclusion Criteria:

* Age Over 40

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: African-American Cased-Based
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-05-12 (Actual)

PRIMARY OUTCOMES:
Questionnaire/Screening | 30 days
  The tool, intended to assess college students' by classmates, includes one portion that is an online self-administered questionnaire. Guidance counselors can use the questionnaire to identify college students students who have been targeted for "Fraud."

CONTACTS AND LOCATIONS:
Locations (1):
- The Southern University, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
Behavioral Analysis- Punishment is the least effective method of changing behavior Causes only a "temporary suppression of the behavior" Behavior returned when punishment discontinued

REFERENCES:
- See also: Related Info — http://www.nih.gov
- See also: Related Info — http://www.subr.edu